CLINICAL TRIAL: NCT03174223
Title: Influence of Deep Versus Moderate Neuromuscular Blockade During General Anesthesia on 30-day Readmission Rates: A Retrospective Analysis of Patient Chart Data
Brief Title: Influence of Deep Versus Moderate Neuromuscular Blockade During General Anesthesia on 30-day Readmission Rates
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Albert Dahan, Clinical Professor, Leiden University Medical Center
Other Study IDs: p17.031
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Complications; Postoperative Wound Infection; Pneumonia
MeSH Terms: conditions — Postoperative Complications; Surgical Wound Infection; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep neuromuscular block: patients received a continuous rocuronium dose to maintain a depth of neuromuscular block of 1-2 twitches post tetanic count
  Interventions: Drug: deep neuromuscular block
- moderate neuromuscular block: patients received neuromuscular block aimed at > 0 twitches train of four

INTERVENTIONS:
Drug: deep neuromuscular block — a continuous dosing of rocuronium is used to achieve neuromuscular block of 1-2 twitches post tetanic count
  Groups: Deep neuromuscular block

SUMMARY:
Deep neuromuscular block (NMB) has shown to produce superior surgical conditions during various abdominal and non abdominal surgeries. It is however unknown if the application of deep NMB leads to favourable outcome, such as lower rate of postoperative complications in general and surgical infections in specific and ultimately lower readmission rates. In the leiden university medical center, deep NMB is routinely applied for a variety of procedures, most notably laparoscopic abdominal and retroperitoneal surgery, eye surgery and neuro radiologic intervention surgery, since 2014. This retrospective study intends to investigate whether the application of deep NMB for these procedures affects patient outcome and readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* deep neuromuscular block
* moderate neuromuscular block
* general anesthesia
* complete anesthesia chart

Exclusion Criteria:

* incomplete anesthesia chart
* missing data regarding postoperative complications or readmission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for laparoscopic abdominal surgery, eye surgery or neuro radiologic intervention surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Readmission | 30 days after surgery
  readmission to the hospital

SECONDARY OUTCOMES:
Cost | 30 days after surgery
  The total cost, including sugammadex use and readmission cost

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands